CLINICAL TRIAL: NCT00952172
Title: Effectiveness of Stair Stepping Exercise Training on Cardiopulmonary Fitness and Sleep Situation in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Stair Stepping Exercise Training in Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chang Gung University, School of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 95-2314-B-182-032-MY3; CGMH-IRB-94-935B
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Sleep Apnea Syndrome
Keywords: Stair stepping training; OSAS; cardiopulmonary fitness; sleep disturbance; Actigraphy
MeSH Terms: conditions — Sleep Apnea Syndromes; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: stair stepping exercise — Stair stepping exercise performed at home daily for eight weeks

SUMMARY:
This 3-year prospective, randomized, control, longitudinal study is aimed to (1) examine the effect of stair stepping exercise training on cardiopulmonary fitness and sleep situation in patients with Obstructive Sleep Apnea Syndrome (OSAS), and (2) follow the longitudinal change after stair stepping exercise training in patients with OSAS. Patients meet the following criteria will be invited to participate in this study: being diagnosed with AHI (Apnea-hypopnea index)>15/hr and ODI (oxygen desaturation index)>10/hr by Polysomnography, aged 19 or older. Based on the power analysis, 70 patients with OSAS treated in the outpatient department of Chang Gung Medical Center will be recruited over a period of 26 months. Each patient will participate in this study for seventeen weeks. Patients will be randomly assigned to receive stair stepping exercise in addition to nursing education and standard care, or nursing education and standard care alone. Stair stepping exercise will be performed at home daily for eight weeks. Outcomes will be determined by changes in the scores of cardiopulmonary fitness index, VO2max, six-minute walking distance, daytime sleepiness measured by Epworth Sleepiness Scale, sleep time measured by Actigraphy, and AHI measured by Polysomnography; those taken four times: before treatment (baseline), five weeks, nine weeks, and seventeen weeks of the study. Data will be analyzed using descriptive statistics and Generalized Estimating Equation (GEE).

DETAILED DESCRIPTION:
This study seeks to verify improvements of the stair stepping exercise training on cardiopulmonary fitness condition and sleep condition in patients with obstructive sleep apnea syndrome (OSAS). The quasi-experimental, two group repeated-measures study design was used. Patients meet the following criteria were invited to participate in this study: being diagnosed with AHI (Apnea-hypopnea index)>15/hr and ODI (oxygen desaturation index)>10/hr by Polysomnography, aged 19 or older. Eighteen patients with OSAS treated in the outpatient department of Chest Medicine were recruited, included study group and control group .The study group patients performed stair stepping exercise training daily for eight weeks at home. Outcome measures included cardiorespiratory fitness condition assessed by the 3-Minute YMCA Step Test, in which including physical fitness index and gross oxygen consumption (VO2), and sleep condition assessed by Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, and Polysomnography. Data were recorded just prior to the stair stepping exercise at Day 1 as baseline, at the end of the fourth week, and at the end of the eighth week. Results of this study showed, physical fitness index, Epworth Sleepiness Scale , AHI, Pittsburgh Sleep Quality Index and symptom scale-snoring were significantly improved. Differences in the effect of stair stepping exercise for other outcome variables were either minimal or not statistically significant. Eight weeks of stair stepping exercise training could be useful in increasing cardiorespiratory fitness condition and improving sleep condition on patients with OSAS.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with AHI (Apnea-hypopnea index)>15/hr and ODI (oxygen desaturation index)>10/hr by Polysomnography
* aged 19 or older

Exclusion Criteria:

* unstable angina

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Hwa Maa, DSN, Principal Investigator — Chang Gung University